CLINICAL TRIAL: NCT07035951
Title: The VIP-3 (Very Old Intensive Care Patients) Study: Decision-making in the Older Intensive Care Unit (ICU) Patient: How Are Family Meetings Implemented Across Diverse Cultures in Europe?
Brief Title: The VIP3 (Very Old Intensive Care Patients) Study: Family Involvement in Treatment Decisions for Old ICU Patients
Acronym: VIP3
Status: Not yet recruiting | Type: Observational
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 337942
Record Dates: First submitted 2025-05-13; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Family Members; Critical Illness; Frailty; Communication; Patient Preference
Keywords: Elderly; Critical illness; communication; frailty; family meetings; Intensive care; critical care; shared decision making; patient preference
MeSH Terms: conditions — Critical Illness; Frailty; Communication; Patient Preference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients age 75 and above admitted as an emergency to Intensive Care: The investigators will be looking at communication whilst these patients are on the Intensive Care Unit (ICU). In particular whether a family meeting takes place (to discuss progress and patient wishes) and if so what is discussed in the meeting.
  In addition to the information taken during the family meeting, the investigators will be collecting the following: baseline demographics, physiological data, frailty score and baseline function, treatments received and outcome data

SUMMARY:
The demographics of the global population is changing with increasing numbers of elderly and co-morbid patients. As a result, more elderly patients will be admitted to the Intensive Care Unit (ICU), which will bring several ethical challenges. It is for this reason the investigators have chosen to focus on this historically neglected and important patient population.

Little is known about how family meetings are implemented in ICUs in Europe and other parts of the world. However, these meetings contribute to building trust between the family and the ICU team. They are a crucial component for planning and conducting a time limited trials as they provide the opportunity for shared-decision making with the ICU team and with other stakeholders.

The investigators plan to determine the current practice of communication between ICU staff and patients and their relatives. The investigators expect to find a substantial variation in approaches to family meetings. This information may then help design and further investigate targeted interventions enabling shared decision-making focused on family and patient values.

The investigators research aim is to to investigate whether Family meetings are used in ICUs across Europe and other regions and, if so, how they are conducted and the influence on patient-centred outcome measures.

DETAILED DESCRIPTION:
This is a prospective observational cohort study in patients aged 75 years old and above admitted as an emergency to the ICU and expected to have a length of stay of 3 days or more.

Consent varies between European countries. In some countries it will be taken on admission, in some (UK) it will be taken after the family meeting or on discharge from ICU and in others it has been waived.

1. information about the study will be given to the patient/consultee and around 24 hours will be allowed for them to have a think about participating or ask the research team any questions
2. If consent has been gained, the research team will record basic demographics of the patient and specific physiological data from the day of admission to the ICU.
3. The research nurse will have a conversation with the patient or next of kin regarding how the patient was prior to admission. If there are no next of kin information will be taken from the notes. From this information, the investigator can determine the clinical frailty scale which will be determined by looking at a proforma and determining which category of frailty the patient best fits. Other baseline information taken will be activities of daily living and co-morbidities.
4. The research nurse will document whether a Family Meeting (FM) takes place, if it does, they will document information about the FM in the electronic CRF. The information will be sought from the patient notes and the doctor or nurse who was in the meeting. If a FM does not take place this will be recorded. In the UK only ,a separate questionnaire about communication on ICU will be given to family members to complete.
5. The outcome of the FM and the patient will be documented
6. survival at 30 days, discharge information and location will be recorded by looking at the hospital records.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Intensive Care Unit (ICU) of participating centres
* Age 75 years and above
* Expected Length of stay (LOS) > 3 days

Exclusion Criteria:

* Refusal to participate
* Limitation of treatment upon ICU arrival (other than Cardiopulmonary Resuscitation-CPR)
* Planned admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Emergency patients admitted to the intensive care unit age 75 years and older. The investigators will ask participating ICUs to include the first consecutive 20 patients or all patients (if <20) admitted within a 6 month period.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a structured/planned family meeting | Until Intensive care unit (ICU) discharge
  The number of patients that have a family meeting during the intensive care stay

SECONDARY OUTCOMES:
Median day since Intensive care unit (ICU) admission when the family meeting took place | Until ICU discharge
  Day number on ICU when family meeting took place
Number of people present in the Family Meeting | Until ICU discharge
  The total number of participants in the family meeting
Categorical description of people present in the Family Meeting | Until ICU discharge
  What were the roles of the participants in the family meeting (patient relatives, doctors, nurses, other health professionals.)
The treatment level after the family meeting | Until ICU discharge
  Treatment level category decided upon at the end of the family meeting which will be either: continuation of care, therapy reduced due to improvement, therapy withheld (WH), therapy withdrawn (WD).
Change in SOFA (Sequential Organ Failure Assessment) score between ICU admission and day of Family Meeting (FM) | Until ICU discharge
  Change in SOFA score from admission to the day of the family meeting. The SOFA score is a tool used to assess the severity of organ dysfunction in a critically ill patient. The total score ranges from 0-24, a higher SOFA score indicates a sicker patient and therefore a worse outcome
Survival until intensive care unit discharge | ICU discharge
  The number of patients that survive to Intensive care unit discharge
Intensive care unit (ICU) length of stay | ICU discharge
  The length of time the participant stays on intensive care (hours)
Hospital survival | From randomisation to hospital discharge, assessed up to 3 months
  The number of participants alive at hospital discharge
Hospital length of stay | From randomisation to hospital discharge, assessed up to 3 months
  The length of time the participant spends in hospital
Discharge location | From randomisation to hospital discharge, assessed up to 3 months
  Where patient is discharged to after discharge from hospital. Is it home, residential home, nursing home or other
Decision to limit life sustaining treatment | Until ICU discharge
  If there is a decision made to withdraw or with hold life sustaining treatment while the patient is on the intensive care unit. This is a yes / no answer
Time between limiting life sustaining treatment and death or ICU discharge | From ICU admission until the first documented progression or date of death from any cause, whichever came first, assessed up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Leaver, PhD FRCP FICM, Principal Investigator — St George's Hospital; Bertrand Guidet, Principal Investigator — l'Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ranzani OT, Besen BAMP, Herridge MS. Focus on the frail and elderly: who should have a trial of ICU treatment? Intensive Care Med. 2020 May;46(5):1030-1032. doi: 10.1007/s00134-020-05963-1. Epub 2020 Mar 2. No abstract available. PMID 32123988
- [Background] Vink EE, Azoulay E, Caplan A, Kompanje EJO, Bakker J. Time-limited trial of intensive care treatment: an overview of current literature. Intensive Care Med. 2018 Sep;44(9):1369-1377. doi: 10.1007/s00134-018-5339-x. Epub 2018 Aug 22. PMID 30136140
- [Background] Beil M, Guidet B, Flaatten H, Jung C, Sviri S, van Heerden PV. Is It TIME for More Research on Time-Limited Trials in Critical Care? Chest. 2022 Jun;161(6):e397. doi: 10.1016/j.chest.2022.01.065. No abstract available. PMID 35680329
- [Background] Chang DW, Neville TH, Parrish J, Ewing L, Rico C, Jara L, Sim D, Tseng CH, van Zyl C, Storms AD, Kamangar N, Liebler JM, Lee MM, Yee HF Jr. Evaluation of Time-Limited Trials Among Critically Ill Patients With Advanced Medical Illnesses and Reduction of Nonbeneficial ICU Treatments. JAMA Intern Med. 2021 Jun 1;181(6):786-794. doi: 10.1001/jamainternmed.2021.1000. PMID 33843946
- [Background] Robinson JD, Jagsi R. Physician-Patient Communication-An Actionable Target for Reducing Overly Aggressive Care Near the End of Life. JAMA Oncol. 2016 Nov 1;2(11):1407-1408. doi: 10.1001/jamaoncol.2016.1948. No abstract available. PMID 27414802
- [Background] Flaatten H, De Lange DW, Morandi A, Andersen FH, Artigas A, Bertolini G, Boumendil A, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zaferidis T, Guidet B; VIP1 study group. The impact of frailty on ICU and 30-day mortality and the level of care in very elderly patients (>/= 80 years). Intensive Care Med. 2017 Dec;43(12):1820-1828. doi: 10.1007/s00134-017-4940-8. Epub 2017 Sep 21. PMID 28936626
- [Background] Guidet B, de Lange DW, Boumendil A, Leaver S, Watson X, Boulanger C, Szczeklik W, Artigas A, Morandi A, Andersen F, Zafeiridis T, Jung C, Moreno R, Walther S, Oeyen S, Schefold JC, Cecconi M, Marsh B, Joannidis M, Nalapko Y, Elhadi M, Fjolner J, Flaatten H; VIP2 study group. The contribution of frailty, cognition, activity of daily life and comorbidities on outcome in acutely admitted patients over 80 years in European ICUs: the VIP2 study. Intensive Care Med. 2020 Jan;46(1):57-69. doi: 10.1007/s00134-019-05853-1. Epub 2019 Nov 29. PMID 31784798
- [Background] Vallet H, Schwarz GL, Flaatten H, de Lange DW, Guidet B, Dechartres A. Mortality of Older Patients Admitted to an ICU: A Systematic Review. Crit Care Med. 2021 Feb 1;49(2):324-334. doi: 10.1097/CCM.0000000000004772. PMID 33332816
- [Background] Guidet B, Leblanc G, Simon T, Woimant M, Quenot JP, Ganansia O, Maignan M, Yordanov Y, Delerme S, Doumenc B, Fartoukh M, Charestan P, Trognon P, Galichon B, Javaud N, Patzak A, Garrouste-Orgeas M, Thomas C, Azerad S, Pateron D, Boumendil A; ICE-CUB 2 Study Network. Effect of Systematic Intensive Care Unit Triage on Long-term Mortality Among Critically Ill Elderly Patients in France: A Randomized Clinical Trial. JAMA. 2017 Oct 17;318(15):1450-1459. doi: 10.1001/jama.2017.13889. PMID 28973065
- [Background] Guidet B, Flaatten H, Boumendil A, Morandi A, Andersen FH, Artigas A, Bertolini G, Cecconi M, Christensen S, Faraldi L, Fjolner J, Jung C, Marsh B, Moreno R, Oeyen S, Ohman CA, Pinto BB, Soliman IW, Szczeklik W, Valentin A, Watson X, Zafeiridis T, De Lange DW; VIP1 study group. Withholding or withdrawing of life-sustaining therapy in older adults (>/= 80 years) admitted to the intensive care unit. Intensive Care Med. 2018 Jul;44(7):1027-1038. doi: 10.1007/s00134-018-5196-7. Epub 2018 May 17. PMID 29774388
- [Background] Bassford C, Griffiths F, Svantesson M, Ryan M, Krucien N, Dale J, Rees S, Rees K, Ignatowicz A, Parsons H, Flowers N, Fritz Z, Perkins G, Quinton S, Symons S, White C, Huang H, Turner J, Brooke M, McCreedy A, Blake C, Slowther A. Developing an intervention around referral and admissions to intensive care: a mixed-methods study. Southampton (UK): NIHR Journals Library; 2019 Nov. Available from http://www.ncbi.nlm.nih.gov/books/NBK549962/ PMID 31765112